CLINICAL TRIAL: NCT02494908
Title: Can Diffusion Tensor MRI Brain Scan Demonstrate Microstructural Changes as Evidence of Neuroplasticity Following a Learning Process in Patients With Idiopathic Parkinson's Disease ?
Brief Title: Evidence of Neuroplasticity After Performing a Cognitive Task in Idiopathic Parkinson's Disease Patients
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Dr. Sharon Hassin (Other Government)
Collaborators: Bar-Ilan University, Israel (Other); Tel Aviv University (Other); Sheba Medical Center (Other Government)
Responsible Party: Sponsor-Investigator, Dr. Sharon Hassin, Dr., Sheba Medical Center
Organization: Sheba Medical Center (Other Government)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: 2372-15-SMC
Record Dates: First submitted 2015-07-08; First posted 2015-07-10 (Estimated); Last update posted 2015-07-10 (Estimated); Status verified 2015-07

CONDITIONS: Parkinson Disease
Keywords: Parkinson Disease; MRI
MeSH Terms: conditions — Parkinson Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Healthy controls (Active Comparator): Healthy controls with no known neurological disease matched for sex and age with the patients group
  Interventions: Behavioral: Playing a computer game simulating a car race
- IPD patients (Active Comparator): Men and women diagnosed with idiopathic parkinson's disease
  Interventions: Behavioral: Playing a computer game simulating a car race

INTERVENTIONS:
Behavioral: Playing a computer game simulating a car race — Playing a computer game simulating a car race

SUMMARY:
As seen in previous studies Diffusion Tensor Imaging (DTI) MRI is able to detect very subtle changes in brain tissue even after a very short timescale of hours resulting from performing a cognitive task and learning, We wish to explore and compare those changes to patients with idiopathic PD (IPD) and see if there are changes in the learning process and can we detect them using widely available noninvasive techniques such as MRI.

DETAILED DESCRIPTION:
Aim: to utilize high sensitivity DTI MRI methodology to explore evidence for subtle microstructural brain alterations after performing a cognitive task and to compare those changes in patients with PD to healthy controls of the same age.

PD patients and controls will undergo a full cranial MRI scan for depiction of anatomy and structural abnormalities (scan duration ~40 min). Immediately afterwards the subjects will play a car race computer game (Need for Speed) for 90 minutes. Following the game, the patients will undergo an additional DTI MRI scan (~15 minutes).

ELIGIBILITY:
Inclusion Criteria:

* Patients with IPD based on a clinical diagnosis of PD according to the United Kingdom Parkinson's Disease Society Brain Bank criteria (however patients with a positive family history and symmetrical onset may be included)
* Healthy subjects should have no known neurological disease matched for age and sex with the study group

Exclusion Criteria:

* History of cranial surgery, radiation therapy, tumor, stroke or significant head trauma
* History of psychiatric disease (major depression, bipolar affective disorder, schizophrenia)
* Patients with severe tremor or dyskinesias that may interfere with performance of the MRI scan
* Patients with Montreal Cognitive Assessment (MoCA) score of 22 or under
* Contraindications for MRI (metal objects: implants/shrapnel/bullet; any electrically, magnetically or mechanically activated implants: cardiac pacemakers/defibrillator, biostimulators, neurostimulators, cochlear implants, hearing aids, insulin pump; claustrophobia)
* Subjects who are familiar and have played on multiple occasions the computer game "need for speed"

Ages: 30 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2015-07; Primary Completion 2018-01 (Estimated); Study Completion 2018-07 (Estimated)

PRIMARY OUTCOMES:
seeing evidence of microstructural brain tissue changes in Diffusion Tensor Imaging (DTI) MRI | 2 hours

CONTACTS AND LOCATIONS:
Overall Officials: Sharon Hassin-Baer, Dr, Principal Investigator — Sheba Medical Center
Locations (1):
- Movement Disorders Institute, Sheba Medical center, Ramat Gan, Israel

REFERENCES:
- [Background] Sagi Y, Tavor I, Hofstetter S, Tzur-Moryosef S, Blumenfeld-Katzir T, Assaf Y. Learning in the fast lane: new insights into neuroplasticity. Neuron. 2012 Mar 22;73(6):1195-203. doi: 10.1016/j.neuron.2012.01.025. Epub 2012 Mar 21. PMID 22445346
- [Background] Vakil E, Herishanu-Naaman S. Declarative and procedural learning in Parkinson's disease patients having tremor or bradykinesia as the predominant symptom. Cortex. 1998 Sep;34(4):611-20. doi: 10.1016/s0010-9452(08)70518-5. PMID 9800094
- [Background] Exner C, Koschack J, Irle E. The differential role of premotor frontal cortex and basal ganglia in motor sequence learning: evidence from focal basal ganglia lesions. Learn Mem. 2002 Nov-Dec;9(6):376-86. doi: 10.1101/lm.48402. PMID 12464697
- [Background] Doyon J, Bellec P, Amsel R, Penhune V, Monchi O, Carrier J, Lehericy S, Benali H. Contributions of the basal ganglia and functionally related brain structures to motor learning. Behav Brain Res. 2009 Apr 12;199(1):61-75. doi: 10.1016/j.bbr.2008.11.012. Epub 2008 Nov 17. PMID 19061920
- [Background] Gheysen F, Van Opstal F, Roggeman C, Van Waelvelde H, Fias W. The neural basis of implicit perceptual sequence learning. Front Hum Neurosci. 2011 Nov 11;5:137. doi: 10.3389/fnhum.2011.00137. eCollection 2011. PMID 22087090
- [Background] Hofstetter S, Tavor I, Tzur Moryosef S, Assaf Y. Short-term learning induces white matter plasticity in the fornix. J Neurosci. 2013 Jul 31;33(31):12844-50. doi: 10.1523/JNEUROSCI.4520-12.2013. PMID 23904619
- [Background] Hill RA. Do short-term changes in white matter structure indicate learning-induced myelin plasticity? J Neurosci. 2013 Dec 11;33(50):19393-5. doi: 10.1523/JNEUROSCI.4122-13.2013. No abstract available. PMID 24336705
- [Background] Foerde K, Shohamy D. The role of the basal ganglia in learning and memory: insight from Parkinson's disease. Neurobiol Learn Mem. 2011 Nov;96(4):624-36. doi: 10.1016/j.nlm.2011.08.006. Epub 2011 Sep 16. PMID 21945835
- [Background] Schlaug G. Musicians and music making as a model for the study of brain plasticity. Prog Brain Res. 2015;217:37-55. doi: 10.1016/bs.pbr.2014.11.020. Epub 2015 Feb 11. PMID 25725909
- [Background] Blumenfeld-Katzir T, Pasternak O, Dagan M, Assaf Y. Diffusion MRI of structural brain plasticity induced by a learning and memory task. PLoS One. 2011;6(6):e20678. doi: 10.1371/journal.pone.0020678. Epub 2011 Jun 20. PMID 21701690